CLINICAL TRIAL: NCT04662853
Title: Gut Microbiota-based Tool for the Detection of Color-rectal Cancer in Positive Patients for the Fecal Occult Blood Test.
Brief Title: Gut Microbiota and Color-rectal Cancer.
Acronym: CCR-microbiota
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Collaborators: Reina Sofia University Hospital (Unknown); Junta de Andalucia (Other Government)
Responsible Party: Sponsor
Other Study IDs: CCR early diagnosis
Record Dates: First submitted 2020-11-19; First posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Cancer; Colo-rectal Cancer; Diagnoses Disease; Microbiota-related Disease; Intestinal Disease
Keywords: Diagnosis improvement; Early diagnosis; Mathematical modelling; Gut microbiota; Colonoscopy
MeSH Terms: conditions — Neoplasms; Colonic Neoplasms; Intestinal Diseases; Disease | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — Feces samples collected before colonoscopy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with positive results in the fecal occult blood test.: Patients with positive results in the fecal occult blood test in the Program for Early Detection of Colon and Rectal Cancer, undergone by the Consejeria de Salud de la Junta de Andalucia (Spain), were invited to participate in the CCR-microbiome study. This program is screening Andalusian population aged between 50 and 69 years old for colo-rectal cancer presence by fecal occult blood test, and further colonoscopy when positive for this test. Patients included in CCR-microbiome study were recruited between January 2017 and March 2020, at the Reina Sofia University Hospital (Cordoba, Spain) with the consumption of antibiotic within the previous month as exclusion criteria.
  Interventions: Diagnostic Test: Gut microbiota determination from feces samples.

INTERVENTIONS:
Diagnostic Test: Gut microbiota determination from feces samples. — Determination of the gut microbiota composition by 16S metagenomic and building of a mathematical model, on the basis of the colonoscopies results, able to classify patients without and with color-rectal cancer-related lessions. These latter will be also classified according to the type of lession.
  Other Names: Colonoscopy

SUMMARY:
This clinical trial is focused in the development of a screening test for the people at risk of colo-rectal cancer (aged more than 50 years old), valid and safe, improving the screening prognosis increasing the sensitivity and sensitive as compared with the current method, fecal occult blood.

DETAILED DESCRIPTION:
Colo-rectal cancer (CCR) is one of the most prevalent cancers in developed countries. Several studies suggest that the CCR may be related with changes in the gut microbiota. This clinical trial is focused in the development of a screening test for the people at risk of CCR (aged more than 50 years old), valid and safe, improving the screening prognosis. The main potential improvement lies in the fact that the proposed method is more specific and sensitive than the current method, fecal occult blood. It aims to distinguish whether the positive results for fecal occult blood test is due to fissures, not related with CCR (which are positive for fecal occult blood, false positive) or was caused by a cancer-related lesion. The methodology derived will also improve the sensitive as sometimes the polyps do not leak blood. Based in the previous differences found in the gut microbiota composition related with CCR for several research groups, the gut microbiota composition will be used as diagnosis tool.

ELIGIBILITY:
Inclusion Criteria:

-Patients with positive results in the fecal occult blood test in the Program for Early Detection of Colon and Rectal Cancer, undergone by the Consejeria de Salud de la Junta de Andalucia (Spain).

Exclusion Criteria:

-The consumption of antibiotic within the previous month to inclusion in the study.

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with positive results in the fecal occult blood test in the Program for Early Detection of Colon and Rectal Cancer, undergone by the Consejeria de Salud de la Junta de Andalucia (Spain), were invited to participate in the CCR-microbiome study. This program is screening Andalusian population aged between 50 and 69 years old for colo-rectal cancer presence by fecal occult blood test, and further colonoscopy when positive for this test. Patients included in CCR-microbiome study were recruited between January 2017 and March 2020, at the Reina Sofia University Hospital (Cordoba, Spain) with the consumption of antibiotic within the previous month as exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Gut-microbiota-based color-rectal cancer diagnosis. | A week before colonoscopy.
  Determination of the gut microbiota composition by 16S metagenomic, data analysis and building of a mathematical model to test the potential use of the gut microbiota architecture as biomarker to color-rectal cancer prognosis in patients with positive results in fecal occult blood test.

SECONDARY OUTCOMES:
Colonoscopy clinical results. | At week 2.
  Prevalence of the different color-rectal cancer lessions.
Characteristic of the population. | A week before colonoscopy.
  The characteristic of the population includes gender (man/woman), age (years), weight in kilograms and height in meters (weight and height will be combined to report BMI in kg/m^2), which will be used to check for any association with the prevalence of the different color-rectal cancer lesions.
Dietary habits | A week before colonoscopy.
  The dietary habits will be assessed by a questionnaire and will be used to check for any association with the prevalence of the different color-rectal cancer lessions.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Hervas, Study Director — Reina Sofia University Hospital; Carmen Haro, PhD, Study Director — Maimonides Institute for Biomedical Research; Antonio Camargo, PhD, Principal Investigator — Maimonides Institute for Biomedical Research
Locations (1):
- Reina Sofia University Hospital, Córdoba, Cordoba, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Microbiota row data.